CLINICAL TRIAL: NCT04342234
Title: Neural Network to Calculate Morphology of the Cleft Palate to Reduce Cleft Lip and Palate Treatment Burden.
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Botnar Research Centre for Child Health (BRCCH) (Unknown); sciCORE Basel (Unknown); Department of Computer Science, Computer Graphics Laboratory, ETH Zurich (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2020-00388; ch19Mueller2
Record Dates: First submitted 2020-04-08; First posted 2020-04-10 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Cleft Palate; Orofacial Cleft
Keywords: Cleft Lip; Neural Network; palatal plate therapy; palatal 3D geometry; palatal shape reconstruction
MeSH Terms: conditions — Cleft Palate; Cleft Lip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: data collection of palatal casts and palatal images of cleft patients routinely treated at the institution — data collection of palatal casts and palatal images of cleft patients, using routinely taken intraoral/palatal photographs and palatal casts of infants with cleft lip and palate deformity

SUMMARY:
This study is to develop a neural network to compute palatal three dimensional (3D) geometry by using routinely taken intraoral/palatal photographs and palatal casts of infants with cleft lip and palate deformity for reducing cleft lip and palate treatment burden. Data of palatal casts and palatal images of cleft patients routinely treated at the University Hospital Basel will be analyzed.The collection of large data helps in developing a neural network that will allow the computation of the 3D geometry from single photographs.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cleft lip and palate malformation with available routinely performed plaster cast model from palatal impressions, intraoral scans from the palate and corresponding images of the cleft palate (1970 till 2025)

Exclusion Criteria:

* Existence of a documented rejection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with cleft lip and palate malformation with available routinely performed plaster cast model from palatal impressions and/or intraoral scans of palate, and corresponding images of the cleft palate treated in the past as well as future patients treated at University hospital Basel (USB) for the last 50 years will be included (1970 till 2025). Models were (until 2020) and intraoral scans are (since 2020) taken routinely in newborns and for follow-up (age 1-20 years) according to WHO Guidelines.
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2020-03-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
3D palatal geometry | at baseline
  palatal cleft photographs (input) and corresponding 3D palatal geometry (output) create this 3D palatal geometry for development of image based, non-invasive palatal shape reconstruction

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Müller, PD Dr. med. Dr. med. dent. Dr., Principal Investigator — Mund-, Kiefer- und Gesichtschirurgie, Universitätsspital Basel
Locations (1):
- Mund-, Kiefer- und Gesichtschirurgie, Universitätsspital Basel, Basel, Switzerland